CLINICAL TRIAL: NCT01599962
Title: Influence of Cincalcet on Cognitive Functions in Healthy Human Subjects
Acronym: Mira-Basel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Director of the Division of Cognitive Neuroscience, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2012DR2027
Record Dates: First submitted 2012-05-02; First posted 2012-05-16 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Memory Functions
MeSH Terms: interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cinacalcet (Experimental)
  Interventions: Drug: Cinacalcet
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Cinacalcet; Drug: Placebo

INTERVENTIONS:
Drug: Cinacalcet — single administration, 90mg
Drug: Placebo — single administration
  Arms: Sugar pill

SUMMARY:
To investigate the effects of the calcimimetic agent cinacalcet on cognitive functions in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* normotensive
* native or fluent German-speaking
* caucasian (European ancestry)
* BMI between 19 and 27 kg/m2

Exclusion Criteria:

* acute or chronic psychiatric or somatic disorder
* pathological ECG
* Low serum calcium
* known hypersensitivity to the IMP
* pregnancy
* breast-feading
* long-term medication within last 3 months
* smoking more than 3 cigarettes per day
* seizures in participants and first degree relatives
* concurrent participation in another study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change of attention functions under cinacalcet | two study days within 10 days
Change of memory functions under cinacalcet | two testing days within 10 days

SECONDARY OUTCOMES:
Change of emotional state under cinacalcet | two study days within 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, Prof. MD, Study Director — University of Basel
Locations (1):
- University of Basel, Division of Cognitive Neuroscience, Basel, Basel, Switzerland